CLINICAL TRIAL: NCT02924103
Title: Danish Title: Afprøvning af indføringsrør Til Forureningsfri Podning af næsens Bihuler (Den Forureningsfri Podepind)
Brief Title: Contamination Free Bacterial Swap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kåre Håkansson (Other)
Collaborators: Region Capital Denmark (Other)
Responsible Party: Sponsor-Investigator, Kåre Håkansson, MD, Ph.D, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CIV-16-04-015264
Record Dates: First submitted 2016-06-06; First posted 2016-10-05 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Sinusitis
Keywords: acute rhinosinusitis; staphylococcus aureus; nasal vestibule; contamination
MeSH Terms: conditions — Sinusitis; Staphylococcal Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right side (Active Comparator): All included participants serve as their own control. A bacterial swab (Eswab 481CE, Copan Diagnostics, Italy), will be introduced to both sides of the nose (to the middle meatus); on the RIGHT side by using the "Contamination free bacterial swab" introduction device.
  The "Contamination free bacterial swab" introduction device is a prototype developed for clinical testing.
  Interventions: Device: Contamination free bacterial swab
- Left side (Active Comparator): All included participants serve as their own control. A bacterial swab (Eswab 481CE, Copan Diagnostics, Italy) will be introduced to both sides of the nose (to the middle meatus); on the LEFT side using the present day clinical procedure (visually guided introduction).
  Interventions: Device: Contamination free bacterial swab

INTERVENTIONS:
Device: Contamination free bacterial swab — A comparison of the bacteriology in bacterial swabs (Eswab 481CE, Copan Diagnostics, Italy) from the middle meatus. On the RIGHT side using the "Contamination free bacterial swab" introduction device that facilitates the introduction of a bacterial swab into the nose without direct or indirect contact with the nasal vestibule.

SUMMARY:
A test of a newly designed device (Contamination free bacterial swab). This device can be used to introduce a standard bacterial swab into the nose without direct or indirect contact with the nasal vestibule.

DETAILED DESCRIPTION:
Aim:

The investigators want to improved the current method for bacterial culture test in patients with possible sinusitis by reducing the risk of contamination from the nasal vestibule. The investigators will examine whether significantly fewer Staphylococcus Aureus are detected in the middle meatus when applying a new device for bacterial swab introduction. This device is designed to prevent bacterial pollution from the nasal vestibule.

More precisely, the investigators hope to reduce the frequency of Staphylococcus aureus in nasal swabs from 10-15 % to 0-5 %.

The overall objective is to avoid over-treatment with broad-spectrum antibiotics in patients with sino-nasal disease.

Design:

A comparative study in which patients serve as their own control. A bacterial swab will be introduced to both sides of the nose; on the right side using the new device, on the left side using the present day technique (visual guidance). 70 participants will be included.

Statistics:

A chi-square test will be used for comparison of frequencies.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of upper airway disease

Exclusion Criteria:

* mental illness
* Need for interpreter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Frequency of staphylococcus aureus positive cultures | 1 year
  Comparison of the frequency of staphylococcus aureus positive cultures from the two sides of the nose

SECONDARY OUTCOMES:
Frequency of other bacteria in cultures | 1 year
  Comparison of the frequency of other positive cultures from the two sides of the nose

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Ørntoft, MD, Principal Investigator — Steffen Ørntoft, Ear, Nose and Throat specialist clinic
Locations (1):
- Ørelæge Steffen Ørntoft, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided